CLINICAL TRIAL: NCT00612066
Title: An Open Label, Multicenter Study Evaluating the Safety and Efficacy of Short Term (6 Weeks) Rosiglitazone Treatment in Patient's With Cushing's Disease
Brief Title: Rosiglitazone in Treating Patients With Newly Diagnosed ACTH-Secreting Pituitary Tumor (Cushing Disease)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual and funding term ended
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000586468; UCLA-0612080-01
Record Dates: First submitted 2008-02-08; First posted 2008-02-11 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2016-01

CONDITIONS: Cushing's Disease
Keywords: ACTH-producing pituitary tumor
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rosiglitazone (Experimental)
  Interventions: Drug: rosiglitazone maleate

INTERVENTIONS:
Drug: rosiglitazone maleate

SUMMARY:
RATIONALE: Rosiglitazone may help pituitary tumor cells become more like normal cells, and to grow and spread more slowly.

PURPOSE: This phase II trial is studying how well rosiglitazone works in treating patients with newly diagnosed ACTH-secreting pituitary tumor (Cushing disease).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effect of rosiglitazone on biochemical control in patients with newly diagnosed ACTH-secreting pituitary tumor (Cushing disease).

Secondary

* To assess the effect of this drug on corticotrophin (CRH)-stimulated pituitary tumor ACTH secretion.
* To assess the overall safety and tolerability of this drug in these patients.
* To assess the overall quality of life of patients treated with this drug.
* Percentage of Reduction in 24-hour Urinary-free Cortisol Levels

OUTLINE: This is a multicenter study.

Patients receive oral rosiglitazone once daily for 7 weeks in the absence of disease progression or unacceptable toxicity.

Blood, urine, and saliva samples are collected periodically for laboratory studies. Inflammatory markers (C-reactive protein, interleukin-6 [IL-6], serum sialic acid, soluble intracellular and vascular adhesion molecules [sICAM-1, and sVCAM-1], and amyloid A) are measured at baseline and at the completion of study treatment; salivary cortisol and 24-hour urinary-free cortisol levels are measured at baseline and weekly during study treatment; dexamethasone suppression tests with serum cortisol and corticotrophin (CRH) stimulation test are performed at baseline and at the completion of study treatment; prolactin, insulin-like growth factor-1 (IGF1), thyroid function, and sex steroid hormones are measured at baseline and at the completion of study treatment; and dynamic pituitary function testing (arginine/growth hormone-releasing hormone [GHRH] testing to measure growth hormone secretion) is performed at baseline.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically demonstrable ACTH-secreting pituitary tumor

  * Pituitary tumor demonstrated on MRI with and without contrast AND/OR evidence of a central ACTH source following inferior petrosal sinus sampling
  * Newly diagnosed disease
* Biochemically active disease that is not adequately controlled, as demonstrated by the following standard criteria:

  * Elevated 24-hour urinary-free cortisol levels on at least 2 separate 24-hour urine collections 1 week apart
  * Lack of suppression of serum cortisol to < 1.8 μg/dL (at 8 am) following administration of 1 mg of dexamethasone at 11 pm the night before
  * Measurable plasma ACTH levels
* Patient is hypercortisolemic and does not wish to receive alternate steroid-lowering therapy, such as ketoconazole and/or metyrapone
* Patients with evidence of optic nerve or chiasm compression on post-operative MRI must have a normal visual field evaluation by Goldman perimetry

  * No visual field abnormalities
* Hypopituitarism* allowed, as evidenced by any or all of the following:

  * Subnormal growth hormone (GH) response to arginine/growth hormone-releasing hormone (GHRH) testing (normal response is an increase of > 4 ng/mL)
  * Low age-and sex-matched insulin-like growth factor-1 (IGF-1) levels
  * Low thyroid-stimulating hormone (TSH) levels
  * Low free triiodothyronine (T3) and free thyroxine (T4) levels
  * Low estradiol levels
  * Low luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in postmenopausal female patients
  * Low testosterone, LH, and FSH levels in male patients NOTE: *Patients who are diagnosed with hypopituitarism will initiate thyroid hormone replacement therapy prior to pituitary surgery as part of routine care. Other hormone replacement, such as sex steroids or growth hormone, will not be initiated during the study.

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception (if oral contraception is used, it must be used for ≥ 2 months prior to, during, and for 1 month after completion of study therapy)
* No clinically significant renal, hematologic, or hepatic abnormalities
* No prior or concurrent medical condition that may interfere with the conduct of the study or the evaluation of its results, in the opinion of the investigator or the DSMB compliance officer
* No history of immunocompromise, including HIV positivity by ELISA and western blot
* No alcohol or drug abuse within the past 6 months
* No blood donation (≥ 400 mL) within the past 2 months
* No other active malignant disease within the past 5 years except for basal cell carcinoma or carcinoma in situ of the cervix
* No active or suspected acute or chronic uncontrolled infection
* No severe osteoporosis, defined as bone mineral density T scores < 2.5 standard deviations below age-matched controls
* No history of noncompliance to medical regimens
* Considered reliable
* Able to complete the entire study

PRIOR CONCURRENT THERAPY:

* More than 3 months since prior rosiglitazone or other thiazolidinedione
* No prior or concurrent radiotherapy for pituitary tumor
* More than 1 month since prior participation in any clinical investigation involving an investigational drug
* More than 30 days since prior unlicensed drugs
* No concurrent pituitary surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Heaney, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period May 2006-May 2009
Groups:
- Rosiglitazone: Rosiglitazone maleate :
Period: Overall Study
Arm/Group | Rosiglitazone
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rosiglitazone
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders
Description: Definition of Treatment Response
  * The primary outcome in Cushing's disease will the % responders, a responder is defined as a patient with 2 consecutive 24h urinary free cortisols within the normal reference range in association with no clinical signs of disease progression.
  * Secondary outcomes will include the % reduction in 24h UFC (derived by comparison of the mean of 2 baseline 24h UFC values with mean of the two lowest consecutive 24h UFC values while on study treatment in association with no clinical signs of disease progression).
Time Frame: 7 weeks
Population: Sample size was too small to do a valid analysis.
Measure: Number; unit: participants
Arm/Group | Rosiglitazone
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Arm/Group | Rosiglitazone
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone (N=2)
edema in limbs (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment was a major limitation. Patients were available but were not interested in the study due to possible side effects of the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No